CLINICAL TRIAL: NCT02378259
Title: AMOS2 (Adolescent Morbid Obesity Surgery)
Brief Title: Randomized Clinical Trial; Medical vs Bariatric Surgery for Adolescents (13-16 y) With Severe Obesity
Acronym: AMOS2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 578-13
Record Dates: First submitted 2014-08-26; First posted 2015-03-04 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Diabetes; Hypertension; Steatohepatitis; Inflammation
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension; Fatty Liver; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomisation between Bariatric surgery (mainly Roux-en-Y gastric bypass) or Intensive Medical treatment
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bariatric surgery (Experimental): Roux-en-Y gastric bypass surgery
  Interventions: Procedure: Laparoscopic Roux-en-Y gastric bypass
- Intense conservative treatment (Active Comparator): Intense conservative treatment. 8 week LCD followed by outpatient visits 1/ month
  Interventions: Procedure: Intense conservative treatment

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-Y gastric bypass — Bariatric surgery with Roux-en-Y gastric bypass as preferred option, possible laparoscopic Vertical Sleeve Gastrectomy
  Arms: Bariatric surgery
Procedure: Intense conservative treatment — Intense medical treatment for obesity (behavioral treatment, dietary intervention, exercise, medication etc) 8 week period of Low Calorie Diet. Treatment intensity about 1 visit a month over 2 years
  Arms: Intense conservative treatment

SUMMARY:
Severe childhood obesity is associated with both immediate and chronic health problems and a severe impact on psychosocial development. Medical and behavioural interventions rarely result in the significant, durable weight loss necessary to improve health outcomes.

This is a randomised clinical trial where 50 adolescents, 13-16 years of age, will be randomised to either early bariatric surgery (Roux-en-Y gastric bypass) or intense conservative treatment and possibly surgery after two years of non-surgical treatment or as they have become 18 years.

DETAILED DESCRIPTION:
A multicentre randomised clinical trial where three tertiary referral hospitals recruit patients.

Patients and their parents receive information about the study at their paediatric clinic and at the trial web page (www.amos2.se). Standardised procedure, including signed informed consent.

Interventions

At the end of day of baseline examination patients are randomised to either of two arms:

* Bariatric surgery with regular follow up
* Optimised conservative treatment starting with an 8-week Low Calorie Diet period followed by tailored support and treatment by the multidisciplinary team with an intensity of at least one visits a month over at least 2 years

Patients in the conservative arm will be reassessed regarding interest of undergoing bariatric surgery two years after inclusion.

Sample Size A sample size of 50 (25+25) leaves a power of more than 95% to evaluate a possible superiority of >10% weight difference between the two groups, assuming a 15% standard deviation in weight loss over follow-up at 2.5% significance level.

This number also allows assessment for differences in cardiovascular risk factors with sufficient power and acceptable power for demonstrating differences in quality of life and cognitive functions.

3.6 Randomization The computerized random allocation is performed during the day of baseline examination and patients were informed of their assignment. Forty-nine patients have been included until May 2017, and the last patient will be operated on June 14th. Stratification has been performed according to the recruitment centre

3.8 Statistical Methods & Additional Analyses Safety & Efficacy Outcomes: Analyses will be by intention to treat, including all randomised patients. Difference in treatment effect will be evaluated with hazard ratio between the treatment groups, and the corresponding confidence interval will be calculated. For secondary outcomes, the incidence of comorbidities during follow-up will be evaluated using time-to-event models, and for continuous variables mixed models will be used to evaluate differences between the treatment groups.

Incremental cost-effectiveness analysis will be conducted by calculating the incremental cost-effectiveness ratio (ICER; dividing the between-group difference in costs with the between-group difference in quality-adjusted life-years (QALYs) as well as life-years). Probabilistic sensitivity analysis will be conducted and results presented in an ICER scatterplot and cost-effectiveness acceptability curve.

Follow-Up Clinical Data Collection: Study point are 6 weeks, 1 year, 2 years, and 5 years after the start of intervention. Weight, quality of life, and adverse events, as well as clinical data regarding treatments for co-morbidities. Blood sampling for assessment of nutritional deficiencies, glucose control, blood lipids and inflammation will be collected at baseline and 1, 2 and 5 years.

Cognitive functions: Assessments will be performed at baseline and 1 and 2 years after start of intervention.

Register-Based Data Collection and Health-Economic Outcomes: Collection and analysis of Swedish national health care and other official registries

We decided in the Study Steering Committee to change time points for long term follow up to be 5, 10 and 15 years after treatment initiation to better comply with standard schedules for clinical follow up in registers (instead of 7, 12 and 17y after treatment initiation).

ELIGIBILITY:
Inclusion Criteria:

* Age 13-16 years
* BMI >35
* Failed comprehensive treatment for obesity > 1 year
* Passing assessment of psychologist
* Tanner 3 or more

Exclusion Criteria:

* Monogenic obesity (for example Prader Willis, Laurence Moon-Bardet-Biedl)
* Obesity secondary to brain injury
* Severely mentally disabled
* Not eligible for general anesthesia
* Psychotic or other major psychiatric illness
* Previous major gastrointestinal surgery

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (kg/m2) | 2 years after treatment initiation

SECONDARY OUTCOMES:
Metabolic control | 2, 5, 10 and 15 years after treatment initiation
  Glucose control (fP-Glc, fs-Insulin, HbA1c, Oral glucose tolerance test), Blood lipids (HDL, LDL, TG, Apo A, Apo B), Blood pressure (systolic and diastolic), Inflammation (LPK, CRP, Adiponectin, IL-6, TNF-alfa), liver function tests (AST, ALT, ALP, Bil)
Quality of life, generic | 2, 5, 10 and 15 years after treatment initiation
  Mental and physical quality of life assessed by Short Form-36 (score 0-100, lower= more disability)
Obesity-specific quality of life | 2, 5, 10 and 15 years after treatment initiation
  Obesity Problem scale- 9 items (score 0-100, higher score= more psychosocial impairment)
Socioeconomic development | 5, 10 and 15 years after treatment initiation
  Education, civil status, number of children, income, sick leave (from national registries)
Health care consumption | 2, 5, 10 and 15 years after treatment initiation
  In hospital care, outpatient care, prescribed medications; from national registries
Skeletal maturation and quality | 2, 5, 10 and 15 years after treatment initiation
  Bone mineral content and bone mineral density will be assessed as well as blood markers for bone formation and resorption
Addictive behavior | 2, 5, 10, 15 years after treatment initiation
  Alcohol consumption, blood markers for alcohol consumption, drugs, brain response to visual stimuli
Mental health | 2, 5, 10 and 15 years after treatment initiation
  Depression, anxiety, self esteem, stability in neuropsychiatric disease (ADHD, ADD), psychiatric illness, OCD
Adverse events | 2, 5, 10 and 15 years after treatment initiation
  Any adverse event (physical, mental or other)
Eating function | 2, 5, 10 and 15 years after treatment initiation
  Assessment of meal pattern, dietary composition and gastrointestinal symptoms in relation to eating
Energy expenditure | 5 years after treatment initiation
  Doubly labelled water, basic metabolic rate, 24h energy expenditure chamber 5 years
Body Mass Index, body weight, height. Additional assessments of primary outcome | 5, 10 and 15 years after treatment initiation
  Weight (kg) and height (m) will be combined to report BMI in kg/m2
Cognitive Function | 1, 2 and 5 years after treatment initiation
  General cognitive functioning (IQ test- WISC-IV Wechsler Intelligence Scale for Children) Scale 1-200 where lower score means worse)
Working memory | 1, 2 and 5 years after treatment initiation
  Memory (D-KEFS-Delis-Kaplan Executive Function System) several subscales 0-15, lower value means worse
Attention | 1, 2 and 5 years after treatment initiation
  Attention (NEPSY- NEuroPSYcologic examination). Separate subscales for executive function and attention, language, memory and learning, sensorimotor, visuospatial processing, and social perception. Lower value means worse.

OTHER OUTCOMES:
Cancer or precancerous lesions | 15 years after treatment initiation and later
  As this parameter is hard to foresee we might need to extend the time for assessment longer than 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Olbers, MD, PhD, Principal Investigator — University of Gothenburg, Dept of Surgical Sciences
Locations (3):
- Sweden (3):
  - Sahlgrenska University hospital, Gothenburg
  - Skåne University Hospital, Malmo
  - Karolinska University hospital, Stockholm

REFERENCES:
- [Derived] Jarvholm K, Gronowitz E, Janson A, Peltonen M, Sjogren L, Beamish AJ, Dahlgren J, Martensson J, Olbers T. Cognitive functioning in adolescents with severe obesity undergoing bariatric surgery or intensive non-surgical treatment in Sweden (AMOS2): a multicentre, open-label, randomised controlled trial. EClinicalMedicine. 2024 Feb 27;70:102505. doi: 10.1016/j.eclinm.2024.102505. eCollection 2024 Apr. PMID 38685922
- [Derived] Jarvholm K, Janson A, Peltonen M, Neovius M, Gronowitz E, Engstrom M, Laurenius A, Beamish AJ, Dahlgren J, Sjogren L, Olbers T. Metabolic and bariatric surgery versus intensive non-surgical treatment for adolescents with severe obesity (AMOS2): a multicentre, randomised, controlled trial in Sweden. Lancet Child Adolesc Health. 2023 Apr;7(4):249-260. doi: 10.1016/S2352-4642(22)00373-X. Epub 2023 Feb 24. PMID 36848922
- [Derived] Janson A, Jarvholm K, Gronowitz E, Sjogren L, Klaesson S, Engstrom M, Peltonen M, Ekbom K, Dahlgren J, Olbers T. A randomized controlled trial comparing intensive non-surgical treatment with bariatric surgery in adolescents aged 13-16 years (AMOS2): Rationale, study design, and patient recruitment. Contemp Clin Trials Commun. 2020 Jun 27;19:100592. doi: 10.1016/j.conctc.2020.100592. eCollection 2020 Sep. PMID 32637723

DOCUMENTS (1):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT02378259/Prot_000.pdf